CLINICAL TRIAL: NCT01584011
Title: Taste Disorders in Middle Ear Disease and After Middle Ear Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: CTN1; CTN12 (Other: UppsalaU)
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-04

CONDITIONS: Taste Disturbance
Keywords: Taste; Chorda tympani nerve
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of nerve tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Middle ear disease
  Interventions: Other: taste measurement; Other: Symptom questionnaire; Behavioral: Quality of life questionnaire; Other: Nerve sample

INTERVENTIONS:
Other: taste measurement — Taste measurements with Electrogustometry and Filter paper test before and after surgery until one year after surgery
Other: Symptom questionnaire — Answering a symptom questionnaire before and after surgery until one year after surgery
Behavioral: Quality of life questionnaire — Answering a quality of life questionnaire before and one year after surgery
Other: Nerve sample — Collect nerve samples from patients undergoing surgery because of vestibular schwannoma, chronic otitis media or cholesteatoma where the nerve cant be saved during planned operation.

SUMMARY:
Objectives

To evaluate the impact of taste disturbance in different types of chronic middle ear diseases and after middle ear surgery.

Hypothesis

That patients with chronic otitis media and cholesteatoma has taste disturbance already before surgery due to the disease itself, of course depending on degree of the disease.

That patients with otosclerosis, has a normal nerve function before surgery.

That patients with normal taste before surgery are more likely to notices a taste disturbance.

That nerve in continuity after surgery, even if it is maltreated, gives less taste disturbance than a divided nerve.

Methods

A clinical study has been launched that measures taste function with two different methods for taste measurements, electrogustometry (EGM) and the filter paper disc method (FPD) before and after middle ear surgery in patients operated with middle ear surgery because of otosclerosis, chronic otitis media and cholesteatoma. The investigators plan to include 120 patients in this study.

A parallel study of the patients own experience of the symptom has also been launched were the patients answer a questionary and a quality of life document. The investigators plan to include 300 patients in this study.

A histological study where specimens of CTN from healthy ears and from ears with chronic disease will be investigated with electron microscopy has also started.

DETAILED DESCRIPTION:
Taste sensations are provided by three different nerves of which the chorda tympani nerve (CTN) is the major taste nerve. It innervates taste buds in the two anterior thirds of the tongue. The CTN location in the middle ear predisposes for trauma of the nerve. In various forms of middle ear pathology, such as chronic otitis and cholesteatoma the nerve can be affected by the pathologic process per se, since the nerve may become exposed to bacteria toxins, enzymes or mechanical damage. During middle ear surgery, it can be cut off, stretched, touched or dried out by the heat of the microscope light beam. The nerve function in these situations is not clarified. Is it for example better to cut the nerve than to leave it traumatized after surgery. Therefore previous reports on objective CTN function pre- and postoperatively unfortunate suffer from inadequate descriptions of ear disease that were studied. In order to elucidate these questions and to give the surgeon deeper knowledge about how to handle CTN during surgery a prospective study is initiated on patients to be operated on with primary middle ear surgery.

We believe that patients with chronic otitis media and cholesteatoma has taste disturbance already before surgery due to the disease itself, of course depending on degree of the disease, and that patients with otosclerosis has a normal nerve function before surgery. We also believe that patients with normal taste before surgery are more likely to notice a taste disturbance and that a nerve in continuity after surgery, even if it is maltreated, gives less taste disturbance than a divided nerve. Two methods of taste measuring are used in the study, Electrogustometry (EGM) and a Filter Paper Disc method (FPD). We have evaluated EGM regarding possible bias and artifacts as well as the correlation regarding results from the two methods.

The study contains three substudies or arms.

1. A clinical prospective trial where 100 patients that undergoes primary middle ear surgery because of chronic otitis, cholesteatoma or otosclerosis are evaluated with EGM and FPD before and after surgery. They also answer a questionnaire about subjective taste disturbance and a questionnaire about quality of life.
2. A clinical multi center study on 200 patients that undergoes primary surgery because of otosclerosis. These patients answer a questionnaire about subjective taste disturbance and a questionnaire about quality of life.
3. A histological study with electron microscopy of CTN from healthy ears and from ears whit chronic otitis or cholesteatoma. We we plan to investigate samples from five healthy and from five sick ears with EM.

ELIGIBILITY:
Inclusion Criteria:

* Patients that undergoes primary middle ear surgery due to chronic otitis media, cholesteatoma and otosclerosis

Exclusion Criteria:

* Not primary surgery
* Not able to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned for primary middle ear surgery due to chronic otitis media, cholesteatoma and otosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Taste disturbance | One year postoperative
  Taste disturbance postoperative will be measured with electrogustometry, filter paper disc methode and symptom questionnaire before surgery and at four times after surgery up till one year poatoperative.

SECONDARY OUTCOMES:
Quality of life | one year
  A quality of life evaluation will be performed before surgery and one year after surgery.
Histopathological changes | At the time of surgery
  Electron microscopy investigation of specimen from healthy ears and from ears with chronic otitis media or cholesteatoma were the nerve could not be saved during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Berling, MD, Principal Investigator — 1Center for Clinical Research, County Council of Västmanland and Uppsala University, Västerås, Sweden
Locations (1):
- Vastmanlands sjukhus ENT department, Västerås, Sweden